CLINICAL TRIAL: NCT02794454
Title: A Randomized, Placebo-controlled, Double-blind Study to Evaluate Efficacy of Investigational Product HeezOn Ultra -1/ HeezOn Ultra-2 on Male Sexual Health
Brief Title: A Study to Evaluate Efficacy of Investigational Product HeezOn Ultra -1/ HeezOn Ultra-2 on Male Sexual Health
Acronym: HeezOn-Ultra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Enovate Biolife Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EB/151005/HZ-U/SD
Record Dates: First submitted 2016-05-31; First posted 2016-06-09 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-06

CONDITIONS: Erectile Dysfunction; Premature Ejaculation
MeSH Terms: conditions — Erectile Dysfunction; Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HeezOn Ultra-1 (Active Comparator): HeezOn Ultra-1 includes ingredients like Shilajit, Galangal, Fenugreek. Dose: 2 capsules daily half an hour before dinner to be taken orally for 21 days.
  Interventions: Other: HeezOn Ultra-1
- HeezOn Ultra-2 (Active Comparator): HeezOn Ultra-2 includes ingredients like Arjuna, Galangal, Fenugreek. Dose: 2 capsules daily half an hour before dinner to be taken orally for 21 days.
  Interventions: Other: HeezOn Ultra-2
- Placebo (Placebo Comparator): Placebo consists of Micro-crystalline Cellulose. Dose: 2 capsules daily half an hour before dinner to be taken orally for 21 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: HeezOn Ultra-1
  Arms: HeezOn Ultra-1
Other: HeezOn Ultra-2
  Arms: HeezOn Ultra-2
Other: Placebo
  Arms: Placebo

SUMMARY:
Sexual function is a part of a normal healthy life and considered to be essential for mental, physical and marital well-being. Any derangement in normal function though is a distressing situation for the individual, is often not reported due to embarrassment or due to social stigma. Sexual disorders in men are categorized according to the stage of sexual response affected in terms of disorders of erectile function, ejaculatory function or libido, albeit there is considerable potential for overlap amongst the disorders. The use of current intervention has many side-effects and has been prohibited in cardiovascular condition and also to be taken with caution with other medical condition.

This has led to the development of multiple alternate therapies which are helpful for a limited number of cases but the major concern for all these therapies is their late onset of action and not having a sustained effect.

DETAILED DESCRIPTION:
Enovate Biolife is trying to improvise further their already marketed product HeezOn® by adding new botanicals thus naming it HeezOn Ultra. HeezOn®has been studied on 148 subjects and has proven to be beneficial for subjects with mild to moderate ED. The previous study fell short to capture the data for subjects who were also suffering from PE and their overall quality of life-related to sexual health. Therefore, the trial is designed to study the speedy and sustained effect of the improvised formula on different aspects of sexual dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

1. Planning to have regular sexual activity (more than twice/ week).
2. Body Mass Index should be ≤ 29 kg/m2.
3. Subjects suffering from erectile dysfunction indicated by SHIMscore ≥ 12 and ≤ 16 for more than 3 months and less than 6 months.

   OR
4. Subjects suffering from predominantly from premature ejaculation as indicated by PEDT score more than 11 for more than 3 months and less than 6 months.
5. Fasting blood sugar ≤ 120 mg/dl.
6. The subjects have to be non-smoker and non-alcoholic.

Exclusion Criteria:

1. Subjects having SHIM score <12 and > 16.
2. Subjects suffering from premature ejaculation predominantly as indicated by PEDT score less than 11.
3. Subjects with major psychiatric disorders or severe systemic disorders
4. Subject having uncontrolled diabetes mellitus and hypertensive on active treatment
5. Subjects having history of male sexual dysfunction more than six months in diabetic subjects.
6. Anatomical deformity of the penis such as severe penile fibrosis or Peyronie's disease or phimosis.
7. Subjects detected with HIV and suffering from AIDS.
8. Has an abnormal thyroid stimulating hormone (TSH) level lower than 30% of lower limit normal or more than 30% of upper limit normal.
9. Has erectile dysfunction caused by neurological or endocrine factors such as hyper-prolactinemia.
10. Subjects with history of major systemic disorders.
11. Subject with history of drug abuse.
12. Subjects using medications known to cause sexual dysfunction (cimetidine, spironolactone, thiazides, adrenergic blockers, antidepressants etc.)
13. Subject has participated in any clinical trial within last 30 days.
14. Subjects not ready to sign the consent & unable to comply the protocol.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in scores of Sexual Health Inventory for Men | Day 0, Day 1, Day 3, Day 14 and Day 28

SECONDARY OUTCOMES:
Sexual Hormone Binding Globulin | Day 0 and Day 14
Free Testosterone | Day 0 and Day 14
Change in scores of Sexual Quality of Life - Male | Day 0, Day 1, Day 3, Day 14 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Patil, M.D., Principal Investigator — Maharashtra Medical Council; Shirish Malde, BHMS, Principal Investigator — Maharashtra Council of Homoeopathy Mumbai

IPD SHARING:
Plan to Share IPD: No